CLINICAL TRIAL: NCT03601299
Title: Back to Basics: Addressing Childhood Obesity Through Traditional Foods in Alaska
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alaska Native Tribal Health Consortium (Other)
Collaborators: Rural Alaska Community Action Program, Inc. (RurAL CAP) (Unknown); University of Alaska Fairbanks (Other); University of Alaska Anchorage (Other); Yukon Kuskokwim Health Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5RO1NRO15417-02
Record Dates: First submitted 2018-06-14; First posted 2018-07-26 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional food arm (Experimental): Traditional food-focused menu
  Interventions: Other: Traditional food
- Non-intervention arm (No Intervention): Standard RurAL CAP menu

INTERVENTIONS:
Other: Traditional food — Increasing traditional food consumption through Head start programs in Alaska
  Arms: Traditional food arm

SUMMARY:
Back to Basics is a mixed-methods intervention trial to reduce the prevalence of obese Alaska Native children by increasing the proportion of nutrient-dense traditional and non-traditional foods consumed, and decreasing consumption of sugar-sweetened beverages (SSBs). This 5-year intervention trial targeting 0-5 year olds is conducted in partnership with Rural Community Action Program, Inc. (RCAP) Head Start (HS), Early Head Start (EHS), and Parents as Teachers (PAT) programs in 12 rural Alaskan communities in the Yukon-Kuskokwim (YK) region, where each site is assigned to either a 9-month nutritional education and meal program intervention or a standard education and meal program repeating annually.

This intervention trial aims to increase consumption of local traditional foods and nutrient-dense non-traditional foods, decrease SSB consumption, and decrease prevalence of obesity in children 3-5 years old by: (1) adjusting the nutritional content of existing meal services provided by RCAP to children ages 3-5 years; (2) providing culturally relevant nutrition education to families of children 0-5 years; (3) developing local and community driven initiatives that provide knowledge and skills and engage families in the gathering and preparing of local traditional foods; and (4) incorporating available and emerging resources (e.g. Fish/Farm-to- Schools) to increase integration of traditional foods into the diet.

Phase 1 involves the collection and analysis of formative and baseline data to help guide the intervention in Phase 2.

Phase 1 includes:

1. Gathering baseline height/weight and food/SSB consumption data previously collected on children ages 0-5 years enrolled in YK RCAP programs.
2. Conducting formative studies in the 12 YK communities to better understand attitudes towards childhood obesity and barriers/enablers to traditional foods consumption
3. Creating/integrating a traditional foods-focused nutrition curriculum into RCAP menu programs in YK communities.

5. Work to expand the "Fish to Schools" and "Farm to Preschool" programs into YK RCAP HS programs.

Phase 2 includes implementing:

1. A physical activity curriculum in HS programs in all communities
2. A traditional food in HS menu program in intervention communities
3. A home-based nutrition program in intervention communities
4. A mechanism to document traditional foods important to each community

ELIGIBILITY:
Inclusion Criteria:

* for the Focus Group Discussions: Consenting Alaska Native residents of the 12 communities involved in the study, aged 18 and over.
* for the intervention study: Upon parental or guardian consent, Alaska Native residents of the 12 communities involved in the study, aged 0-5 years and enrolled in the RurAL CAP Head start, Early Head start, or Parents as Teachers, programs

Exclusion Criteria:

* None

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | Measured annually over 4 years of intervention
  Change in Proportion of AN children 3-5 years old with a BMI greater than or equal to the 95th percentile
Traditional food content | Measured annually over 4 years of intervention
  Change in Percentage of total calories derived from traditional foods

CONTACTS AND LOCATIONS:
Overall Officials: Timothy K Thomas, MD, Principal Investigator — Alaska Native Tribal Health Consortium; Kathy Koller, PhD, Study Director — Alaska Native Tribal Health Consortium
Locations (1):
- Alaska Native Tribal Health Consortium, Anchorage, Alaska, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ohle KA, Koller KR, Walch AK, Lee FR, Palmer L, Nu J, Thomas TK. Alaska Native Parents' Decision-Making About Food, Beverages, and Screen Time for Young Children: Formative Insights From the "Got Neqpiaq?" Project. Fam Community Health. 2023 Oct-Dec 01;46(4):250-258. doi: 10.1097/FCH.0000000000000370. PMID 37703513
- [Derived] Hill CM, Paschall MJ, Koller KR, Day GM, Lee FR, O'Brien DM, King DK, Palmer L, Thomas TK, Bersamin A. Obesity Prevalence and Dietary Factors Among Preschool-Aged Head Start Children in Remote Alaska Native Communities: Baseline Data from the "Got Neqpiaq?" Study. Child Obes. 2023 Oct;19(7):498-506. doi: 10.1089/chi.2022.0143. Epub 2022 Dec 5. PMID 36473164
- [Derived] Koller KR, Flanagan CA, Nu J, Lee FR, Desnoyers C, Walch A, Alexie L, Bersamin A, Thomas TK. Storekeeper perspectives on improving dietary intake in 12 rural remote western Alaska communities: the "Got Neqpiaq?" project. Int J Circumpolar Health. 2021 Jan 1;80(1):1961393. doi: 10.1080/22423982.2021.1961393. PMID 34350814